CLINICAL TRIAL: NCT01318616
Title: The Effect of Strength Training on the Hip Adduction Strength Measured With Hand-held Dynamometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amager Hospital (Other)
Responsible Party: Principal Investigator, Kristian Thorborg, phd, Amager Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: H-4-2010-119
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Hip Adduction Strength
Keywords: hip adduction strength training; Improvement in adductor strength

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Training group (Experimental)
  Interventions: Other: Strength training of the hip adductors

INTERVENTIONS:
Other: Strength training of the hip adductors — Adductor strength training

SUMMARY:
The purpose of this study is to investigate the effect of strength training with elastic bands on hip strength in soccer players, the effect measured with hand-held dynamometry. The primary outcomes are isometric and eccentric hip adduction strength. The hypothesis is that strength training with elastic bands will result in a clinical relevant increase in hip adduction strength.

ELIGIBILITY:
Inclusion Criteria:

* Sub-elite danish soccer players

Exclusion Criteria:

* Injury in the lower back or legs with a duration of more than 6 weeks within the last year before the study was initiated.
* Systematic strength training of the hip adductors more than once a week within the last 6 months before the study was initiated.
* Groin pain during soccer play with a duration of more than 1 week and witch resulted in loss of soccer training/game within the last 3 months before the study was initiated.
* Groin injuries within the last month before the study was initiated.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Isometric hip adduction strength | 8 weeks
Eccentric hip adduction strength | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Amager Hospital, Copenhagen, Denmark